CLINICAL TRIAL: NCT01256502
Title: The SERI® Surgical Scaffold Use in Reconstruction Post Market Study for Tissue Support and Repair in Breast Reconstruction Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sofregen Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SURE-001
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Breast Reconstruction

ARMS (1):
- Implanted Participants (Other): Participants with breast reconstruction surgery implanted with SERI® Surgical Scaffold.
  Interventions: Device: SERI® Surgical Scaffold

INTERVENTIONS:
Device: SERI® Surgical Scaffold — Breast reconstruction surgery

SUMMARY:
The purpose of the study is to obtain clinical experience with the use of SERI® Surgical Scaffold for tissue support and repair in breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for enrollment, the subject must:

* Be female, greater or equal to 18 years of age
* Be willing to undergo breast reconstruction with sub-pectoralis muscle placement of a tissue expander, followed by exchange with a sub-pectoral breast implant
* Have previously had or be willing to undergo mastectomy with healthy, well-vascularized skin flaps anticipated by the surgeon
* Be in good health other than breast pathology and be suited to general anesthesia and planned treatments.

Exclusion Criteria:

The subject must not:

* Have undergone breast radiation treatment and/or is preoperatively evaluated to require radiation treatment to the breast area during the course of the study
* Have a known allergy to silk
* Have collagen-vascular, connective disease, or bleeding disorders
* Have a Body Mass Index (BMI) that is greater than or equal to 35
* Have any disease, including uncontrolled diabetes, which is clinically known to impact wound healing ability
* Have an autoimmune disease, an immune deficiency, or is on immune suppression drugs other than any other current treatment for breast cancer
* Have smoked within the last 12 months
* Currently have an alcohol/substance abuse problem or have had a relapse within 1 year prior to screening visit
* Be pregnant, lactating, or expecting to be within the next 24 months
* Have concomitant unrelated condition of breast/chest wall/skin
* Have an abscess or infection at the time of surgery
* Have undergone previous breast surgery with the exception of mastectomy, breast biopsy, cyst removal, lumpectomy, mastopexy, reduction and/or augmentation
* Have had a prior soft tissue support device implanted in the breast
* Have a condition or be in a situation that, in the Investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Allergan Medical
Locations (1):
- Los Angeles, California, United States

REFERENCES:
- [Derived] Fine NA, Lehfeldt M, Gross JE, Downey S, Kind GM, Duda G, Kulber D, Horan R, Ippolito J, Jewell M. SERI surgical scaffold, prospective clinical trial of a silk-derived biological scaffold in two-stage breast reconstruction: 1-year data. Plast Reconstr Surg. 2015 Feb;135(2):339-351. doi: 10.1097/PRS.0000000000000987. PMID 25502862

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment was defined as having signed the IRB-approved Informed Consent Form. 160 patients were enrolled, of which 139 were implanted with SERI® Surgical Scaffold.
Period: Overall Study
Arm/Group | Implanted Participants
Started | 139 (Implanted with SERI during Stage I breast reconstruction surgery)
Completed | 129
Not Completed | 10
Not completed — Had scaffold removed | 4
Not completed — Personal reasons | 5
Not completed — Protocol deviation | 1

BASELINE CHARACTERISTICS:
Population: Subjects implanted with SERI® during their Stage I breast reconstruction surgery
Arm/Group | Implanted Participants
Number analyzed (Participants) | 139
Age, Customized [Number; unit: participants]
  18 to 19 years | 0
  20 to 29 years | 4
  30 to 39 years | 15
  40 to 49 years | 54
  50 to 59 years | 40
  60 to 69 years | 22
  70+ years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 139

OUTCOME MEASURES:

1. Primary Outcome: Investigator Satisfaction Following Use of SERI® Surgical Scaffold at 6 Months
Description: The primary outcome measure was investigator satisfaction at 6 months after stage I surgery/implantation of SERI® Surgical Scaffold. Satisfaction was evaluated using an 11-point scale, where 0=very dissatisfied to 10=very satisfied.
Time Frame: 6 months
Population: Of the 139 participants, 214 breasts, implanted with SERI® during Stage I breast reconstruction, 4 discontinued the study and 1 missed the 6-month visit, leaving 134 subjects, 205 breasts in the primary analysis population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Implanted Participants
Number analyzed (Participants) | 134
units on a scale | 9.4 (0.84)

2. Secondary Outcome: Investigator Ease of Use Assessment at the Time of SERI® Placement During Stage I Surgery
Description: Ease of Use assessments of SERI® Surgical Scaffold by the investigator were collected on Case Report Forms (CRFs) following stage I surgery. Ease of Use was assessed separately using a 5-point scale, where 0=very difficult to 5=very easy to use for the following criteria: • SERI® preparation before implantation (excluding cutting or shaping) • SERI® cutting and shaping before implantation • SERI® positioning/drapability during implantation • SERI® cutting and shaping after implantation • SERI® suturing during implantation (including tension and stretch). The number of participants who were implanted with SERI® Surgical Scaffold (n=139) by Investigator Ease of Use response for each category is reported.
Time Frame: Immediately following Stage I surgery
Population: Full analysis population included all enrolled participants who had SERI® Placement during Stage I Surgery.
Measure: Number; unit: participants
Arm/Group | Very Difficult to Use | Difficult to Use | Neither Difficult Nor Easy to Use | Easy to Use | Very Easy to Use
Number analyzed (Participants) | 139 | 139 | 139 | 139 | 139
participants
  SERI® preparation before implantation | 0 | 0 | 0 | 15 | 124
  SERI® cutting and shaping before implantation | 0 | 0 | 0 | 18 | 121
  SERI® positioning/drapability during implantation | 0 | 0 | 2 | 61 | 76
  SERI® cutting and shaping after implantation | 0 | 0 | 0 | 47 | 92
  SERI® suturing during implantation | 0 | 0 | 1 | 53 | 85

3. Secondary Outcome: Investigator Satisfaction Following Use of SERI® Surgical Scaffold at Other Time Points
Description: Investigator satisfaction with SERI® Surgical Scaffold was evaluated at Stage II surgery and Months 12, 18 and 24 after surgery/implantation using an 11-point scale, where 0=very dissatisfied to 10=very satisfied.
Time Frame: Stage 2 Surgery, Months 12, 18 and 24
Population: Participants from the Full Analysis population (139 participants, 214 breasts), all enrolled participants who had SERI® Surgical Scaffold surgery/implant, with data at the given time-point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Implanted Participants
Number analyzed (Participants) | 134
units on a scale
  Stage 2 Surgery (n=202 breasts) | 9.3 (1.25) [9.06 to 9.47]
  Month 12 (n=198 breasts) | 9.5 (0.89) [9.34 to 9.62]
  Month 18 (n=199 breasts) | 9.4 (1.26) [9.13 to 9.56]
  Month 24 (n=195 breasts) | 9.5 (1.01) [9.41 to 9.72]

ADVERSE EVENTS:
Time Frame: Up to 24 months following SERI implantation
Description: All Serious Adverse Events (SAEs) are reported. All Adverse Events (AEs) occurring at >5% frequency are reported. Individual participants can experience more than 1 AE.
Arm/Group | Implanted Participants
Serious Adverse Events (participants affected / at risk) | 25/139
Other Adverse Events (participants affected / at risk) | 107/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Implanted Participants (N=139)
Cellulitis (Infections and infestations) | 5
Device related infection (Infections and infestations) | 2
Seroma (Injury, poisoning and procedural complications) | 1
Breast cellulitis (Infections and infestations) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Pneumonia (Infections and infestations) | 2
Lobular breast carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Deep vein thrombosis (Vascular disorders) | 1 — This event was classified as unrelated to the SERI® surgical scaffold but related to the surgical procedure. The subject was treated with antihistamines and anticoagulants. The event was reported as serious and ongoing
Pharyngitis (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Vaginal cellulitis (Infections and infestations) | 1
Vaginal ulceration (Reproductive system and breast disorders) | 1 — This event was classified as unrelated to the SERI® surgical scaffold or the procedure and resolved without sequelae after treatment with antipruritics and antibiotics
Parotitis (Infections and infestations) | 1
Salivary gland calculus (Gastrointestinal disorders) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — This event was classified as unrelated to the SERI® surgical scaffold or the procedure. This event remains ongoing.
Atrial fibrillation (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Pericarditis constrictive (Cardiac disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Capsular contracture associated with breast implant (General disorders) | 3
Implant site reaction (General disorders) | 1
Mastitis (Infections and infestations) | 2
Postoperative wound infection (Infections and infestations) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hemiparesis (Nervous system disorders) | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Implanted Participants (N=139)
Procedural pain (Injury, poisoning and procedural complications) | 19
Nausea (Gastrointestinal disorders) | 7
Breast complication associated with device (General disorders) | 12
Capsular contracture associated with breast implant (General disorders) | 10
Seroma (Injury, poisoning and procedural complications) | 13
Wound dehiscence (Injury, poisoning and procedural complications) | 9
Insomnia (Psychiatric disorders) | 9
Erythema (Skin and subcutaneous tissue disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 10
Skin necrosis (Skin and subcutaneous tissue disorders) | 12
Hematoma (Vascular disorders) | 9

LIMITATIONS AND CAVEATS:
None to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As this study involves multiple centers, no individual publications will be allowed prior to completion of the final report of the multicenter study except as agreed with Allergan.